CLINICAL TRIAL: NCT06905847
Title: Phase I Clinical Trial to Evaluate the Safety, Tolerability, Pharmacokinetic and Pharmacodynamics Characteristics of HSK39004 Suspension for Inhalation.
Brief Title: Phase I Clinical Trial to Evaluate the Safety, Tolerability, Pharmacokinetic Characteristics, and Primary Efficacy of HSK39004 Suspension for Inhalation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Haisco Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HSK39004-101
Record Dates: First submitted 2024-12-31; First posted 2025-04-02 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2024-12

CONDITIONS: Healthy Donors

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- HSK39004 in healthy volenteers (Experimental): Single or multiple inhaled HSK39004
  Interventions: Drug: HSK39004 in healthy
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: HSK39004
- HSK39004 in COPD patients (Experimental): multiple inhaled HSK39004
  Interventions: Drug: HSK39004 in COPD

INTERVENTIONS:
Drug: HSK39004 in healthy — 1.5-12mg
  Arms: HSK39004 in healthy volenteers
Drug: HSK39004 — Placebo
  Arms: Placebo
Drug: HSK39004 in COPD — 1.5-6mg
  Arms: HSK39004 in COPD patients

SUMMARY:
To evaluate the safety, tolerability and pharmacokinetic characteristics of HSK39004 suspension for inhalation in single/multiple administration(s) in healthy subjects; to evaluate the safety,tolerability and efficacy of HSK39004 suspension for inhalation in multiple administrations in patients with Chronic Obstructive Pulmonary Disease（COPD）.

ELIGIBILITY:
Inclusion Criteria:

* For healthy volenteers:

  1. Voluntarily sign the informed consent form, understand the trialprocedures, and be willing to comply with all trial procedures andrestrictions;
  2. 18 years to 45 years (inclusive), male and female;
  3. Male subjects weight ≥50 kg and female subjects weight ≥45 kg. Body mass index (BMI) : 18-26 kg/m2 (inclusive) ;
  4. Ability to perform acceptable and reproducible spirometry;
  5. Normal lung function during the screening period, no airway obstruction, FEV1 and forced vital capacity(FVC) are at least 80% of the predicted values;
  6. Subjects are willing to voluntarily use effectivecontraceptives from screening to at least 3 months after the last dose administration.
* For COPD patients:

  1. Voluntarily sign the informed consent form, understand the trialprocedures, and be willing to comply with all trial procedures andrestrictions;
  2. Age ≥ 40 years , male and female;
  3. According to the diagnostic criteria of 2024 Practical Edition of Guidelines , the patient was diagnosed with COPD; The patient has chronic respiratory symptoms such as shortness of breath, chronic cough or expectoration, and/or a history of exposure to risk factors, and the results of pulmonary function tests show that post-bronchodilator spirometry demonstrate FEV1/FVC ratio of ≤0.70 ;
  4. At screening: post-bronchodilator spirometry demonstrate FEV1/FVC ratio of ≤0.70 and FEV1 must be ≥40 % to ≤80% of predicted normal and FEV1 increased by ≥100ml compared with pre-bronchiectasis;
  5. No regular treatment of COPD was performed before joining the study. COPD agents (except SABA and/or SAMA) that are contraindicated in the protocol may be discontinued during the screening and treatment;
  6. Subjects are willing to voluntarily use effectivecontraceptives from screening to at least 3 months after the last dose administration.

Exclusion Criteria:

* For healthy volenteers:

  1. Have a history of severe and uncontrolled diseases, such ascardiovascular, respiratory, liver, gastrointestinal, endocrine,hematologic, mental/nervous systems diseases within 3 months prior to screening;
  2. Have a history of any malignant tumors;
  3. Normal or abnormal vital signs, physical examination, laboratory examination, electrocardiogram, and imageological examination have no clinical significance (only for healthy subjects);
  4. Previous or current gastrointestinal, liver, kidney, or other disease known to interfere with drug absorption, distribution, metabolism, or excretion;
  5. Acute respiratory infections occurred within 6 weeks before screening and/or before randomization;
  6. Have a history of high consumption of grapefruit juice, methylxanthinerich food or beverage (such as coffee, tea, cola, chocolate, energydrinks) ,consumption of grapefruit juice, methylxanthine-rich food within 48 hours before the administration;
  7. Smoking more than 5 cigarettes per day within 3 months prior toscreening or smoking during the study (only for healthy subjects);
  8. Average alcohol intake is more than 14 unit per week (1unit=10g alcohol , 1 unit=285 mL 4.9% alcohol beer, or 30 mL 40% alcohol spirit, or 100mL 12% alcohol wine) within the 3 months prior to screening;
  9. Have a history of drug abuse prior to screening, or positive urine drug screen at screening (If COPD patients were false positives due to other medications, they can be retested after the medication is washed);
  10. Blood donation (or blood loss) ≥400 mL within 3 months prior to the screening;
  11. Subjects who have a allergic to any component of HSK39004 or allergic history to opiates;
  12. Intolerance to this product or the same target drug;
  13. Subjects who use any live vaccine within 30 days prior to screening;
  14. Have participated in any clinical investigator within 3 months prior to screening;
  15. A pregnant/lactating woman, or has a positive pregnancy test at screening or during the trial;
  16. Not suitable for this study as judged by the investigator.
* For COPD patients, in addition to meeting the above exclusion criteria, they should also:

  1. Present with any of the following diseases: Alpha-1 antitrypsin deficiency, asthma, active pulmonary tuberculosis, lung cancer, pulmonary edema, cystic fibrosis, bronchiolitis obliterans, sarcoidosis (sarcoidosis), bronchiectasis, unstable sleep apnea, Or clinically significant pulmonary fibrosis, pulmonary hypertension, or interstitial lung disease determined by the study physician to be a safety risk to the patient and/or to affect the analysis of the study results;
  2. Previous or current history of serious cardiovascular disease;
  3. Have type 1 diabetes or poorly controlled type 2 diabetes (fasting blood glucose ≥10 mmol/L at screening);
  4. During the screening period, the investigators determined that the patient's laboratory tests had clinically significant abnormalities that could pose a safety risk to the patient;
  5. Patients who were hospitalized for COPD or infectious pneumonia within 8 weeks prior to screening and/or had acute exacerbations of COPD or infectious pneumonia between the screening period and prior to randomization, indicating the presence of an active infection;
  6. Patients with acute exacerbations of moderate to severe COPD ≥2 times/year within 1 year before screening;
  7. Acute exacerbations of COPD requiring treatment with oral or parenteral corticosteroids occurred within 8 weeks prior to screening;
  8. Had lung volume reduction surgery within 1 year prior to lung resection or screening;
  9. Patients who use oxygen therapy for long-trem and more than 12 hours per day;
  10. Not suitable for this study as judged by the investigator.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 63 (Actual)
Dates: Start 2024-09-02 (Actual); Primary Completion 2025-01-13 (Actual); Study Completion 2025-03-20 (Actual)

PRIMARY OUTCOMES:
adverse events | From the enrollment of the subjects to 72 hours after the last administration
  The Incidence of adverse events as assessed by CTCAE v5.0

SECONDARY OUTCOMES:
AUC | from 0 to 72 hours after administration
  area under the concentration-time curve
Cmax | from 0 to 72 hours after administration
  maximum plasma concentration
t1/2 | from 0 to 72 hours after administration
  half-life
Vz/F | from 0 to 72 hours after administration
  apparent volume of distribution
CL/F | from 0 to 72 hours after administration
  apparent clearance
Forced Expiratory Volume in the first second (FEV1) for patients with COPD | From 0 before first administration to 24 hours after last administration
  Mean Change From Baseline in Peak FEV1, Mean Change From Baseline FEV1 to Morning Trough FEV1

CONTACTS AND LOCATIONS:
Locations (1):
- West China Hospital of Sichuan University, Chengdu, Sichuan, China